CLINICAL TRIAL: NCT04992091
Title: Constructive Debriefing
Brief Title: Effects of Constructive Debriefing on Procedural Skills and Satisfaction of Nursing Students in Low Fidelity Context. A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Bushra Sultan, Bushra Sultan, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB# 264-754-2019
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Procedural Skill. Learning
Keywords: Debriefing, Procedural skills, Satisfaction, Reflection, Critical thinking
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONSTRUCTIVE DEBRIEFING (Experimental): interventional group
  Interventions: Other: constructive debriefing
- traditional debriefing (No Intervention): noninterventional group

INTERVENTIONS:
Other: constructive debriefing — Constructive debriefing was applied to an interventional group Traditional debriefing was applied on noninterventional group
  Other Names: traditional debrieifng
  Arms: CONSTRUCTIVE DEBRIEFING

SUMMARY:
Purposes: This study was set out to measure the effectiveness of constructive debriefing on procedural skills and satisfaction of nursing students in the low-fidelity context in comparison to traditional debriefing.

Method: The randomized controlled (Parallel double blinded) trial design was used.

Participant: Out of 51 approached, 34 students were selected from the list of participants by a data collector using simple random sampling technique. Following, block randomization was applied using Microsoft Excel to create two equivalent (n=17) groups i.e. experimental and non-experimental.

Setting: The study was conducted in private college of nursing Islamabad Pakistan Intervention: The experimental group received constructive debriefing and non-experimental group received the traditional debriefing. The data were collected using suctioning, sterile dressing skills checklist, and debriefing reflection subscale of Satisfaction with Simulation Experience Scale.

ELIGIBILITY:
Inclusion Criteria:

- Students who were enrolled in the Adult Health Nursing (AHN) course were included in the study

Exclusion Criteria:

* Studentsnts who were repeating the course and were absent for two or more days during skills demonstration and signing off were excluded

Ages: 20 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
learning scores | 8months
  learning scores of participant

SECONDARY OUTCOMES:
satisfaction level | 8months
  measure satisfaction level of participant

CONTACTS AND LOCATIONS:
Locations (1):
- Bushra, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided